CLINICAL TRIAL: NCT06870357
Title: A Study of the Correlation Between the Debilitating State of the Elderly and Propofol Sensitivity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: yuewei20240110
Record Dates: First submitted 2024-11-19; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-01

CONDITIONS: Frailty; Telomere
Keywords: telomere length; propofol; Frailty
MeSH Terms: conditions — Frailty | interventions — Propofol; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- frail group (Experimental): Edmonton scores three or more points
  Interventions: Drug: propofol
- non-frail group (Experimental): Edmonton scores zero to three
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Fifteen minutes after the subarachnoid block, propofol was pumped in at a rate of 20 mg/kg/h with a micro pump, and the pumping rate was reduced to 10 mg/kg/h after 1 min. The infusion was stopped when the consciousness disappeared, and the time of the disappearance of consciousness was observed (time of the disappearance of eyelash reflex).
  Other Names: Ropivacaine

SUMMARY:
In an aging society, there is a surge in the number of surgeries for elderly patients in hospitals, and the elderly are at greater risk of anesthesia due to their own characteristics: slowing metabolism, decreasing resistance, and decreasing physical function, and increased sensitivity to propofol. However, there are large individual differences, and anesthesiologists have found that they cannot judge a patient's sensitivity to anesthetic drugs based on age alone. Patients with different levels of debilitation have different sensitivities to propofol. The use of measuring telomere length to assess the debilitating state of the elderly is a novel and reliable assessment method. Then the sensitivity to propofol of people with different debilitating states was studied, so as to guide anesthesiologists to use drugs safely and reasonably, with a view to realizing the purpose of precise anesthesia.

DETAILED DESCRIPTION:
Part I: A study of the correlation between telomere length and somatic debilitation status in older adults Telomere length was measured by fluorescent quantitative PCR, and subjects were assessed for somatic frailty using the Edmonton Scale (EFS).

1. Perform a correlation analysis between telomere length and Edmonton debility score.
2. Comparison of telomere length differences between Edmonton debility subgroups.
3. Subjects were categorized into "not debilitated" and "debilitated" dichotomous variables according to Edmonton debilitation ratings. The strength of the predictive power of telomere length for frailty was determined using the area under the ROC curve (AUC) using the operator operating characteristic curve ROC treatment .

Part II: Correlation between telomere length and propofol sensitivity in elderly surgical patients A total of 128 patients undergoing lower limb surgery under subarachnoid block in the Second Hospital of Shanxi Medical University were selected and divided into non-frailty group and frailty group.Propofol was pumped at a rate of 20 mg/kg/h with a micropump at 15 minutes after subarachnoid block, and the pumping rate was reduced to 10 mg/kg/h after 1 minute.Stop the infusion when consciousness is absent and observe the time of loss of consciousness (time of loss of eyelash reflex).

intraoperative recording of the time of loss of consciousness (time of disappearance of eyelash reflex), time of awakening, and dosage of propofol in both groups; recording of the time of admission to the room (T0), the time after completion of subarachnoid blockade (T1), the time after 1min of pumping propofol (T2), the time after 5min of pumping propofol (T3), the time after 10min of pumping propofol (T4), the time after 15min of pumping propofol ( T5), after pumping propofol for 20 min (T6), after pumping propofol for 25 min (T7), and after pumping propofol for 30 min (T8); mean arterial pressure (MAP), heart rate (HR), and electroencephalographic dual-frequency index (BIS value) at nine time points; the incidence of adverse reactions (hypotension, bradycardia, and respiratory depression) was recorded for the two groups.

Research hypotheses:

1. There is a difference in propofol sensitivity indices between the debilitated and non-debilitated groups. [time to loss of consciousness; heart rate; MAP; BIS; occurrence of adverse effects; use of vasoactive drugs].
2. There was a difference in telomere length between the debilitated and non-debilitated groups.
3. Among all patients, those with shorter telomere lengths were more sensitive to propofol, and the patients' sensitivity to propofol could be predicted by their telomere lengths.

experimental procedure

1. Comparison of demographic information between the two groups
2. Comparison of propofol sensitivity between the two groups
3. Comparison of telomere length between the two groups.
4. To analyze the correlation between telomere length and its demographic and clinical characteristics for the two groups, the multiple linear regression model was further used to analyze the factors associated with telomere length for all patients, taking the independent variables of gender, age, BMI and other demographic information, and the dependent variable of telomere length. Again, it is shown that there is no significant linear relationship between patients' demographic information and telomere length. Then explain how factors that have a linear correlation will affect the patient's sensitivity to propofol.
5. Analyze the correlation between telomere length and propofol sensitivity indexes, and then use linear regression model to further regress telomere length on the indexes with correlation. The independent variable was selected as telomere length and the dependent variable was time to loss of consciousness/heart rate/MAP/BIS. the model was subjected to analysis of variance (ANOVA) to obtain the β and P values, which indicated whether the model was statistically significant and whether the telomere length could predict several of the above indexes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* American Society of Anesthesiologists (ASA) Classification I-IV
* No previous history of central nervous system disease, no history of psychiatric disorders, no contraindications to anesthesia
* No use of sedative drugs or opioids within 24h
* Approval and consent by the Ethics Committee of Shanxi Medical University and written informed consent by the patient (or authorized delegate)

Exclusion Criteria:

* leukemia patient
* Patients with hearing and visual impairments, communication disorders, inability to complete the debilitating state test
* Patient or family refused to participate in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
telomere length | 24 hours
  Differences in telomere length
Loss of consciousness time | 24 hours
  Differences in loss of consciousness time
awakening time | 24 hours
  Differences in awakening time
Propofol dosage | 24 hours
  Differences in Propofol dosage
Mean Arterial Pressure (MAP) | 24 hours
  Differences in Mean Arterial Pressure (MAP)
heart rate | 24 hours
  Differences in heart rate
Electroencephalographic dual frequency index (BIS value) | 24 hours
  Differences in Electroencephalographic dual frequency index (BIS value)
Incidence of adverse effects (hypotension, bradycardia, respiratory depression) | 24 hours
  Incidence of adverse effects (hypotension, bradycardia, respiratory depression)

SECONDARY OUTCOMES:
Use of vasoactive drugs | 24 hours
  Use of vasoactive drugs

OTHER OUTCOMES:
Checklist form: Sex, age, ASA classification, smoking history, drinking history, comorbidities | 24 hours
BMI | 24 hours
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China